CLINICAL TRIAL: NCT05225896
Title: Clinical-immunological Features of DNER Ataxia
Acronym: CLIMDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 497
Record Dates: First submitted 2022-01-25; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: DNER Ataxia
Keywords: DNER antibodies; autoimmune cerebellar ataxia; Hodgkin lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood and tumors collected at diagnosis time
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DNER ataxia: Patients with well-characterized DNER antibodies.
  Interventions: Genetic: Description of clinical characteristic and genetic tumors

INTERVENTIONS:
Genetic: Description of clinical characteristic and genetic tumors — This is a non-interventional study involving clinical data and biological samples (DNA). Clinical data are collected for the center and samples are already stored in biobank repositories and collected as part of "good clinical practice" in the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population. Patients have already gave explicit written consent for biological specimens sampling and storage at the "Centre de Ressources Biologiques des Hospices Civils de Lyon" (CRB-HCL) (including tissue, cells or biological fluids) and genetic analysis for research purposes. Additionally, patients will be informed about the present study.

SUMMARY:
Using a retrospective cohort of 34 patients with DNER ataxia, we will characterize clinical presentation, tumor associations, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Patient with neurological disorder
* Patient with DNER antibodies in sera or CSF

Exclusion Criteria:

* - No available clinical data
* Patient without DNER antibodies or neurological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with DNER antibodies
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale (mRS) | 6 month after the beginning of study
  Residual neurological disability as assessed by the modified Rankin scale (mRS) score at last visit)

CONTACTS AND LOCATIONS:
Locations (1):
- HCL Hôpital Neurologique / Groupement EST, Bron, France